CLINICAL TRIAL: NCT04999683
Title: Effect of Anti-inflammatory (ITIS) Diet in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Monica Guma, Associate Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 161474
Record Dates: First submitted 2021-08-02; First posted 2021-08-11 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ITIS diet (Experimental): anti-inflammatory (ITIS) diet for 14 days
  Interventions: Dietary Supplement: ITIS diet

INTERVENTIONS:
Dietary Supplement: ITIS diet — anti-inflammatory diet for 14 days

SUMMARY:
to study the effect of anti-inflammatory diet on clinical and biological outcomes in rheumatoid arthritis

DETAILED DESCRIPTION:
The investigators would like to evaluate how inflammation occurs in the joints of subjects with arthritis, and identify molecules and bacteria that can predict whether a rheumatic subject will flare. Blood, urine and stool will be evaluated in the laboratory and compared to their own samples after changes in diet. This is an exploratory study, which is meant to gather preliminary data about the quick effects of changes in diet and treatment on molecules in blood/urine and bacteria in stools. These studies can provide clues to the cause of disease and might ultimately lead to new therapies.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed of rheumatoid arthritis
* without changes in treatment in the last 3 months

Exclusion Criteria:

* food allergies
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change of baseline pain measured by visual analogue scale (0-10) after two weeks of ITIS diet | 2 weeks
  Change of baseline pain measured by visual analogue scale after two weeks of ITIS diet, being 0 no pain, and 10 worse pain

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sala-Climent M, Lal E, Cedola F, Alharthi M, Fernandez-Bustamante M, Agustin-Perez M, Singh A, Choi SI, Rivera T, Nguyen K, Lee S, Golshan S, Holt T, Quehenberger O, Coras R, Guma M. Oxylipin serum profile changes in response to an open-label anti-inflammatory dietary intervention. Clin Nutr ESPEN. 2025 Aug;68:389-402. doi: 10.1016/j.clnesp.2025.05.027. Epub 2025 May 23. PMID 40414498